CLINICAL TRIAL: NCT03296579
Title: A Prospective Open Randomized Clinical Trial of Non-invasive Ventilation Versus Standard Therapy for Children Hospitalized With an Acute Exacerbation of Asthma.
Brief Title: Non-invasive Ventilation vs. Standard Therapy for Children Hospitalized With an Acute Exacerbation of Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Michael Seear, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H17-02008
Record Dates: First submitted 2017-09-21; First posted 2017-09-28 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Asthma Acute; Asthma in Children
MeSH Terms: interventions — Continuous Positive Airway Pressure; Ipratropium; Magnesium Sulfate; Aminophylline; Oxygen; Health Services Needs and Demand

STUDY DESIGN:
Masking Description: It is not possible to use non-invasive face masks on the control patients so the study is unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional asthma therapy. (Active Comparator): Bilevel Positive Airway Pressure group(BiPAP). BiPAP settings at 15/5 cm H2O by face mask with background rate 10 to 15/min. Standard steroid dose plus hourly salbutamol and oxygen to keep SaO2 > 92%.
  Interventions: Drug: Ipratropium; Drug: Magnesium Sulfate; Drug: Aminophylline; Drug: Standard steroid dose, hourly salbutamol, oxygen as needed
- Non-invasive ventilation (CPAP). (Experimental): Continuous Positive Airway Pressure group (CPAP). CPAP settings at 8 to 10 cm H2O. Standard steroid dose plus hourly salbutamol and oxygen to keep SaO2 > 92%.
  Interventions: Device: CPAP; Drug: Standard steroid dose, hourly salbutamol, oxygen as needed
- Non-invasive ventilation (BiPAP) (Experimental): Standard steroid dose, hourly salbutamol, oxygen as needed, nebulized ipratropium q 6 hrly, magnesium sulfate 50 mg/kg IV (4 doses q 6 hrly), loading dose of aminophylline 6 mg/kg IV if no progress.
  Interventions: Device: BiPAP; Drug: Standard steroid dose, hourly salbutamol, oxygen as needed

INTERVENTIONS:
Device: BiPAP — The patient's breathing is assisted by cycling between high and low pressures at a pre-set rate.
  Other Names: Trilogy BiPAP; Bilevel Positive Airway Pressure
  Arms: Non-invasive ventilation (BiPAP)
Device: CPAP — The patient breathes against a constant pressure delivered by face mask.
  Other Names: Continuous Positive Airway Pressure
  Arms: Non-invasive ventilation (CPAP).
Drug: Ipratropium — Nebulized q6h
  Arms: Conventional asthma therapy.
Drug: Magnesium Sulfate — 50mg/kg IV, 4 doses q6h
  Arms: Conventional asthma therapy.
Drug: Aminophylline — 6mg/kg IV (if no progress)
  Arms: Conventional asthma therapy.
Drug: Standard steroid dose, hourly salbutamol, oxygen as needed — Standard common therapies for all three arms.

SUMMARY:
Acute asthma produces greatly increased work of breathing and increased oxygen requirement secondary to bronchial narrowing and airway obstruction by inflammatory secretions. There is growing evidence that non-invasive ventilation can reverse these processes more efficiently than conventional asthma therapy. Surprisingly, there have not yet been any large scale prospective controlled studies to investigate this hypothesis, (either in adults or children). Consequently, the aim of this study is to determine if the use of non-invasive positive airway pressure, for children admitted to hospital with an acute exacerbation of asthma, reduces their work of breathing, need for adjunctive medications, and shortens the length of hospital stay, compared to current standard therapy.

DETAILED DESCRIPTION:
The aim of the study is to determine if the use of NIV, for children admitted to hospital with an acute exacerbation of asthma, reduces their work of breathing, need for adjunctive medication, length of hospital stay, and need for intubation and mechanical ventilation. Study design will be prospective, randomized and controlled. The tightly fitting face mask necessary for NIV makes it impossible to make this a blinded study.

The principal enrollment criteria will be children over 2 years of age presenting to the ER with acute asthma. After diagnosis, all children are treated with standard therapy (systemic steroids plus 3 doses of inhaled salbutamol and 1 dose of inhaled ipratropium over a 1 hour period then hourly salbutamol). The principal decision between discharge track and admission track will be made at 2 hours after first steroid dose. Admission criteria are based on sequential PRAM scores.

After initial asthma treatment and observation in the emergency room, to determine which patients can be discharged home, those who need admission will be asked to join the study, then consented and randomized. There will be three treatment groups:

* BiPAP: standard steroid dose, hourly salbutamol and BiPAP at 15/5 cm H2O by face mask with rate 10 to 15/min, oxygen as needed.
* CPAP: standard steroid dose, hourly salbutamol and 8 to 10 cm H2O constant pressure by face mask, oxygen as needed.
* Conventional therapy: standard steroid dose plus hourly nebulized salbutamol, nebulized ipratropium q 6 hrly, magnesium sulphate 50 mg/kg IV (4 doses q 6 hrly), loading dose of aminophylline 6 mg/kg IV if no progress, oxygen as needed.

All children will be admitted to a small 3 bed respiratory unit. They will be closely monitored and objectively scored every 4 hours using the PRAM asthma clinical severity score (Pediatric Respiratory Assessment Measure). Projected patient enrollment will be at least 30 in each arm. Estimated study duration is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 2-18 years old
* Clinical diagnosis of acute asthma exacerbation (respiratory rate greater than WHO's age-dependent criteria, a history of similar previous episodes and wheezing heard on auscultation by an experienced physician)
* PRAM score of 8 or more after 2 hours post-steroid administration
* Parents willing and able to sign consent
* Children over the age of 6 willing to provide assent

Exclusion Criteria:

* Clinical suspicion of bacterial pneumonia: focal crackles or bronchial breathing, and/or major chest x-ray findings.
* Impending respiratory failure at presentation requiring direct PICU admission
* Any contraindication to BiPAP use including altered mental status, recent bowel surgery, intractable vomiting, inability to protect airway, pneumothorax.
* Receiving maintenance dose of oral steroid at time of hospital admission
* History of serious unrelated illness such as congenital heart disease or bronchopulmonary dysplasia.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Time to reach a PRAM score of ≤3 | Patients will be followed for the duration of their hospital stay (an estimated average duration of 4 days)
  PRAM score includes assessment of oxygen saturations, suprasternal retractions, scalene muscle contraction, air entry and wheezing.

SECONDARY OUTCOMES:
Time to room air | Patients will be followed for the duration of their hospital stay (an estimated average of 4 days).
  Time that oxygen is required
Total medication use per 12 hr period | Patients will be followed for the duration of their hospital stay (an estimated average of 4 days).
  Comparison of total medication use by children in each arm.
Numbers failing treatment and transferred to ICU | Patients will be followed for the duration of their hospital stay (an estimated average of 4 days).
  Number of patients in each group that fail treatment and require transfer to ICU

OTHER OUTCOMES:
Time to reach FEV1 >80% predicted in those children able to perform pulmonary function tests | Patients will be followed for the duration of their hospital stay (an estimated average of 4 days).
  Standard pulmonary function tests can usually be performed by children >6 years.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seear, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gowraiah V, Awasthi S, Kapoor R, Sahana D, Venkatesh P, Gangadhar B, Awasthi A, Verma A, Pai N, Seear M. Can we distinguish pneumonia from wheezy diseases in tachypnoeic children under low-resource conditions? A prospective observational study in four Indian hospitals. Arch Dis Child. 2014 Oct;99(10):899-906. doi: 10.1136/archdischild-2013-305740. Epub 2014 Jun 12. PMID 24925892
- [Background] Basnet S, Mander G, Andoh J, Klaska H, Verhulst S, Koirala J. Safety, efficacy, and tolerability of early initiation of noninvasive positive pressure ventilation in pediatric patients admitted with status asthmaticus: a pilot study. Pediatr Crit Care Med. 2012 Jul;13(4):393-8. doi: 10.1097/PCC.0b013e318238b07a. PMID 22067982
- [Background] Ducharme FM, Chalut D, Plotnick L, Savdie C, Kudirka D, Zhang X, Meng L, McGillivray D. The Pediatric Respiratory Assessment Measure: a valid clinical score for assessing acute asthma severity from toddlers to teenagers. J Pediatr. 2008 Apr;152(4):476-80, 480.e1. doi: 10.1016/j.jpeds.2007.08.034. Epub 2007 Oct 31. PMID 18346499
- [Background] Martinez FD, Vercelli D. Asthma. Lancet. 2013 Oct 19;382(9901):1360-72. doi: 10.1016/S0140-6736(13)61536-6. Epub 2013 Sep 13. PMID 24041942
- [Background] Nava S, Hill N. Non-invasive ventilation in acute respiratory failure. Lancet. 2009 Jul 18;374(9685):250-9. doi: 10.1016/S0140-6736(09)60496-7. PMID 19616722
- [Background] British Thoracic Society Standards of Care Committee. Non-invasive ventilation in acute respiratory failure. Thorax. 2002 Mar;57(3):192-211. doi: 10.1136/thorax.57.3.192. No abstract available. PMID 11867822
- [Background] Nievas IF, Anand KJ. Severe acute asthma exacerbation in children: a stepwise approach for escalating therapy in a pediatric intensive care unit. J Pediatr Pharmacol Ther. 2013 Apr;18(2):88-104. doi: 10.5863/1551-6776-18.2.88. PMID 23798903
- [Background] Papiris SA, Manali ED, Kolilekas L, Triantafillidou C, Tsangaris I. Acute severe asthma: new approaches to assessment and treatment. Drugs. 2009;69(17):2363-91. doi: 10.2165/11319930-000000000-00000. PMID 19911854
- [Background] Green E, Jain P, Bernoth M. Noninvasive ventilation for acute exacerbations of asthma: A systematic review of the literature. Aust Crit Care. 2017 Nov;30(6):289-297. doi: 10.1016/j.aucc.2017.01.003. Epub 2017 Jan 27. PMID 28139368
- [Background] Soroksky A, Klinowski E, Ilgyev E, Mizrachi A, Miller A, Ben Yehuda TM, Shpirer I, Leonov Y. Noninvasive positive pressure ventilation in acute asthmatic attack. Eur Respir Rev. 2010 Mar;19(115):39-45. doi: 10.1183/09059180.00006109. PMID 20956164

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT03296579/Prot_SAP_004.pdf
  • Informed Consent Form (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT03296579/ICF_005.pdf